CLINICAL TRIAL: NCT04154254
Title: Applying PET/MR for Dementia Applications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-19-ES-0586-CTIL
Record Dates: First submitted 2019-10-29; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dementia Patients (Experimental)
  Interventions: Diagnostic Test: PET/MR

INTERVENTIONS:
Diagnostic Test: PET/MR — The PET will be performed with one of the following tracers: 18F-FDG, 18F-DOPA or 18F-flutemetamol (Vizamyl). Proper tracer will be determined by the physician according to the condition. Patients that will agree, will be asked to perform two scans each with different tracer. The 3 tesla magnet of the MRI should allow acquisition of several contrasts within a reasonable time frame. The protocol will include T1 and T2-weighted images, perfusion and diffusion images. Images will be analyzed visually and quantitatively. Quantitative analysis will include MR parameters such as DWI apparent diffusion coefficient (ADC) and PET quantitative metabolic data such as standard uptake values (SUV), metabolic tumor volume (MTV), and total lesion glycolysis (TLG). Hidden image parameters will also be extracted for texture analysis purposes. Quantitative data will be correlated to clinical and pathological data to check accuracy, specificity and sensitivity.

SUMMARY:
Dementia is a common disorder affecting about 50 million people worldwide with nearly 10 million cases every year . It is characterized by cognitive impairments as well as behavior disabilities. Cognitive impairments include difficulties with memory, attention, language and other higher cortical functions. Behavior disabilities may include apathy, aggressive behavior, hallucinations and changes in social interaction. The most common cause of dementia is Alzheimer disease (AD). To plan a proper treatment for the patient it is critical to evaluate accurately the type of dementia as well as obtain the earliest diagnosis possible. However, accurate differential diagnosis in dementia poses difficulties due overlapping phenotypes and limited understanding of the mechanism and pathologies . Diagnosis of the dementia is performed based on the combination of clinical symptoms and biomarkers that include imaging, genetic biomarkers, cerebrospinal fluid (CSF), and other objective markers of disease . The two main modalities used for dementia imaging are Magnetic Resonance Imaging (MRI) and molecular imaging including Single Photon Emission Tomography (SPECT) and Positron Emission Tomography (PET). MRI is performed with various of contrasts such as high resolution T1- weighted, T2- weighted and Diffusion Tensor Imaging (DTI) and functional MRI (fMRI) [2]. These methods give information about morphological modifications in the brain and atrophy characterizing the specific dementia type. In addition brain perfusion and diffusion pattern and assessment of the changing un the resting state functional connectivity network of the brain can be studied with MRI. PET with different tracer molecules allow diagnosis of metabolism pattern in the brain (18F-FDG-PET), modifications in the neurotransmitter system and detection of brain plaques associated with dementia such as amyloid β or Tau aggregates . Data acquired from both modalities allow the reliable and differential diagnosis, prediction of pre-dementia stages, monitoring therapy response and additional research information regarding the mechanism of the condition.

DETAILED DESCRIPTION:
Simultaneous measurements of PET and MR together as is recently became possible have allow spatial and temporal correlation between the two modalities opening a window of opportunities that was not available so far. The first practical advantage is because most neurological patients should go through both MRI and PET scans. Allowing both scans in the occasion significantly increase patient comfort. Furthermore, the simultaneous scans in contrast to sequential scans allow correlation between PET and MR informaiton without the concern of pathological brain modifications between the scans. Currently PET is performed combined with CT, which is superior to MR in the field of brain images. MR high soft tissue resolution as well as extra information it may provide regarding brain perfusion, diffusion, metabolic parameters etc., make the MR a far better modality for brain imaging than CT. In addition, the combined tool allow leveraging MR data to improve PET data quantification. PET issues such as motion correction, partial volume effect and correct localization of the tracer in the brain anatomy that cause PET image degradation and lower accuracy and robustness of PET quantitative parameters, can be solved by integrating MR data into the analysis. Several recently published articles have demonstrated different correction approaches for motion correction and partial volume effect showing an improvement in the PET images both visually and quantitatively . PET attenuation correction using MR data have also been studied, however this matter still need to be resolved. PET/MR for neurological conditions, in general, and specifically for conditions resulting in dementia, is a promising application with a large variety of research opportunities and its abilities need to be explored. Optimization of the acquisition protocols and even more so, the analysis and quantification protocols still need to be performed and will be the focus of this study.

ELIGIBILITY:
Inclusion Criteria:

patients over the age of 18 with diagnosed conditions that might result in dementia or with diagnosed dementia in different stages.

Exclusion Criteria:

1. Patients younger than 18 years
2. pregnancy
3. contraindication to MRI or to intravenous gadolinium injection.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-10 (Estimated); Primary Completion 2021-03-10 (Estimated); Study Completion 2022-01-10 (Estimated)

PRIMARY OUTCOMES:
Patients who preformed PET/MR for dementia applications | 1 year
  Optimization of brain acquisition protocols and reconstruction (with focus on attenuation correction algorithm) for patients with conditions causing dementia.

IPD SHARING:
Plan to Share IPD: Undecided